CLINICAL TRIAL: NCT00002933
Title: CWRU 1296: Biochemical and Pharmacokinetic Predictors of Colon Cancer Response to a Topoisomerase I Directed Treatment With Irinotecan
Brief Title: Irinotecan in Treating Patients With Metastatic or Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: James K.V. Willson, MD, Ireland Cancer Center at University Hospitals Case Medical Center,Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1296
Record Dates: First submitted 1999-11-01; First posted 2004-08-12 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irinotecan hydrochloride — Irinotecan IV at a starting dose weekly for 4 weeks followed by 2 weeks of rest. Treatment continues in the absence of disease progression or unacceptable toxicity. Tumor status is reassessed every 12 weeks during study. Patients attaining a complete response may receive additional courses of treatment. Patients are followed until death.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have metastatic or recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Confirm the greater than 20% response rate to irinotecan in patients with metastatic or recurrent colorectal cancer who have not receive prior chemotherapy for their advanced disease. II. Characterize pharmacokinetic parameters of irinotecan and its metabolite SN-38 and their relationship to response and toxic effect. III. Characterize tumor samples for topoisomerase I activity, proliferative fraction (ki67 expression), and p53 expression and determine whether clinical response is related to these tumor characteristics in patient population. IV. Determine the in vitro inhibition of topoisomerase I activity by irinotecan, SN-38, and other camptothecin analogs and evaluate whether the degree of in vitro sensitivity to irinotecan and/or SN-38 is associated with clinical response in these patients. VII. Determine the frequency of somatic mutations following irinotecan and correlate this with pharmacologic parameters.

OUTLINE: Patients receive irinotecan IV at a starting dose weekly for 4 weeks followed by 2 weeks of rest. Treatment continues in the absence of disease progression or unacceptable toxicity. Tumor status is reassessed every 12 weeks during study. Patients attaining a complete response may receive additional courses of treatment. Patients are followed until death.

PROJECTED ACCRUAL: A total of 54 patients will be accrued into this study at a rate of 25 patients per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or recurrent adenocarcinoma of the colon or rectum that is incurable by surgery or radiation therapy A metastatic lesion in the liver or lung should be evaluated for definitive surgical treatment before being considered for this study Measurable disease required Elevated CEA, hepatomegaly ascites, pleural effusion, positive nuclear scan or bone scan, or poorly defined pelvic or abdominal mass are NOT considered measurable disease Must have measurable disease outside the radiation port or progression of disease within a previously radiated area Must be eligible for a biopsy of a malignant lesion No ascites that are detectable on physical exam No brain metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Greater than 12 weeks Hematopoietic: WBC at least 4,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.2 mg/dL SGOT less than 4 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL or Creatinine clearance at least 60 mL/min Other: No history of any other malignancy except curatively treated nonmelanoma skin cancer and carcinoma in situ of the cervix No active infection or other serious medical conditions deemed unacceptable Negative pregnancy test Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for advanced disease Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy Surgery: At least 3 weeks since any surgical procedure

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1996-09; Primary Completion 2000-07 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of irinotecan in treating patients who have metastatic or recurrent colorectal cancer. | Starting dose weekly for 4 weeks followed by 2 weeks of rest. Treatment continues in the absence of disease progression or unacceptable toxicity. Tumor status is reassessed every 12 weeks during study.

CONTACTS AND LOCATIONS:
Overall Officials: James KV Willson, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio